CLINICAL TRIAL: NCT02181985
Title: A Phase IIIb, Randomised, Open Label Trial With 3 Parallel Groups: Full Dose TNK-tPA Together With Heparin Sodium, Full Dose TNK-tPA Together With Enoxaparin, and Half Dose TNK-tPA Together With Abciximab and Heparin Sodium in Patients With Acute Myocardial Infarction: ASSENT 3 (Assessment of the Safety and Efficacy of New Thrombolytic Regimens)
Brief Title: Full Dose Tenecteplase (TNK-tPA) Together With Heparin Sodium, Full Dose Tenecteplase With Enoxaparin, Half Dose Tenecteplase Together With Abciximab and Heparin Sodium in Patients With Acute Myocardial Infarction (AMI)
Acronym: ASSENT 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123.10
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Heparin; Enoxaparin; Abciximab

ARMS (3):
- TNK-tPA + heparin (Active Comparator)
  Interventions: Drug: Full dose TNK-tPA; Drug: Heparin
- TNK-tPA + enoxaparin (Experimental)
  Interventions: Drug: Full dose TNK-tPA; Drug: Enoxaparin
- TNK-tPA + abciximab + heparin (Experimental)
  Interventions: Drug: Half dose TNK-tPA; Drug: Heparin; Drug: Abciximab

INTERVENTIONS:
Drug: Full dose TNK-tPA
  Arms: TNK-tPA + enoxaparin; TNK-tPA + heparin
Drug: Half dose TNK-tPA
  Arms: TNK-tPA + abciximab + heparin
Drug: Heparin
  Arms: TNK-tPA + abciximab + heparin; TNK-tPA + heparin
Drug: Enoxaparin
  Arms: TNK-tPA + enoxaparin
Drug: Abciximab
  Arms: TNK-tPA + abciximab + heparin

SUMMARY:
The objective of ASSENT 3 was to evaluate the safety and efficacy of full dose tenecteplase with heparin sodium (group A), full dose tenecteplase combined with enoxaparin (group B) and half dose tenecteplase combined with abciximab and heparin sodium (group C).

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms of AMI within six hours prior to randomisation
* A twelve-lead electrocardiogram with one of the following: ST-segment elevation ≥ 0.1 millivolt (mV) in two or more limb leads, or ≥ 0.2 mV in two or more contiguous precordial leads indicative of AMI, or left bundle-branch block
* Age ≥ 18
* Informed consent received

Exclusion Criteria:

* Hypertension defined as blood pressure > 180/110 mm Hg (systolic BP >180 mm Hg and/or diastolic BP >110 mm Hg) on repeated measurements during current admission prior to randomization
* Use of abciximab (ReoPro ®) or other glycoprotein-IIb/IIIa antagonists within the preceding 7 days
* Major surgery, biopsy of a parenchymal organ, or significant trauma within 2 months
* Any minor head trauma and any other trauma occurring after onset of the current myocardial infarction
* Any known history of stroke or transient ischemic attack or dementia
* Any known structural damage of the central nervous system
* Prolonged cardiopulmonary resuscitation (>10 minutes) in the previous two weeks
* Current oral anticoagulation
* Standard unfractionated heparin (heparin sodium) >5000 IU or a subcutaneous dose within 6 hours of randomization of a therapeutic dose of any low molecular weight heparin
* Known thrombocytopenia (prior platelet count below 100000 cells/μl (100 x10**9/l))
* Known renal insufficiency (prior S-creatinine >2.5 mg% (>220 μmol/l) for men and >2.0 mg% (>175 μmol/l)) for women
* Pregnancy or lactation, parturition within the previous 30 days. Women of childbearing potential must have a negative pregnancy test, or use a medically accepted method of birth control
* Treatment with an investigational drug under another study protocol in the past 7 days
* Previous enrollment in this study
* Known sensitivity to TNK-tPA, tPA, abciximab, heparin or low molecular weight heparin
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated
* Inability to follow protocol and comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5989 (Actual)
Dates: Start 2000-05; Primary Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Composite endpoint: 30-day mortality or in-hospital reinfarction or in-hospital refractory ischemia or in-hospital intracranial hemorrhage (ICH) or in-hospital major bleedings (other than ICH) | Up to 30 days after discharge from hospital
Composite endpoints: 30-day mortality or in-hospital reinfarction or in-hospital refractory ischemia | Up to 30 days after discharge from hospital